CLINICAL TRIAL: NCT04444596
Title: Conjunctival Swab vs Nasopharyngeal Swab in Patients With COVID-19
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1104/2020
Record Dates: First submitted 2020-06-18; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-04

CONDITIONS: COVID-19; SARS-CoV 2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Swab (Other): Conjunctival swab and nasopharyngeal swab for SARS-COV 2
  Interventions: Diagnostic Test: Conjunctival swab and nasopharyngeal swab

INTERVENTIONS:
Diagnostic Test: Conjunctival swab and nasopharyngeal swab — Both conjunctival swab and nasopharyngeal swab for SARS-COV 2 are conducted in patients with COVID-19.

SUMMARY:
The aim of this possible study is to identify if SARS-CoV-2 can be found in the tear film and conjunctiva of a patient with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* A confirmed COVID-19 disease
* Signed and dated declaration of consent
* The patient fell ill in Tyrol

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2021-03-31 (Estimated); Study Completion 2021-03-31 (Estimated)

PRIMARY OUTCOMES:
SARS-CoV2 positive conjunctival swabs | 1 year
  The primary endpoint is the number of conjunctival swabs tested positive for SARS-CoV2.

SECONDARY OUTCOMES:
Conjunctival swab vs nasopharyngeal swab | 1 year
  The secondary target is the difference between the conjunctival swab tested positive for SARS-CoV2 and the nasopharyngeal swab.

OTHER OUTCOMES:
Viability of SARS-COV 2 | 1 year
  In the case of a SARS-COV 2 positive conjunctival swab a virus culture will be conducted to clarify, whether it is a viable virus or virus RNA fragments.

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No